CLINICAL TRIAL: NCT03488615
Title: Analyse de la Prise en Charge et de l'Orientation Des Patients de 75 Ans et Plus Consultant Pour Chute Aux Urgences du CHU Angers : données de l'évaluation Initiale et du Recueil de données effectué un an après Leur Passage Aux Urgences
Brief Title: Older falleRs : From Emergency to Geriatric Network
Acronym: OREGoN
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-05
Record Dates: First submitted 2018-01-26; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Fall Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The fall is a complex process associated with high morbidity and mortality, with an institutionalization rate of up to 40% and a major socio-economic impact.

The prevalence of falls increases with age. In fact, it is estimated that one-third of people over 65 and 50% of those over 80 living at home fall at least once a year, half of whom fall repeatedly.

For all these reasons, the fall is a frequent reason for emergency consultation, and is an integral part of geriatric syndromes at risk of early readmission.

The care of the elderly patient has been the subject of good practice recommendations by the Health Authority (HAS) in 2009, with the aim of referring patients to specialized geriatric care. Among these recommendations is the need to look for signs of geriatric severity of falls.

To our knowledge, few studies have investigated the applicability of HAS recommendations with the practice of emergencies; this study is part of a project to improve practices.

- Hypothesis : Due to the fast pace of emergency medicine, the complexity of elderly patients and the inherent limitations of the care system, we hypothesize that few serious fallers are included in the geriatric pathway after admission to the emergency room (ER).

DETAILED DESCRIPTION:
From the database of URQUAL software available at the Emergencies of Angers Hospital and the "list of diagnostics for clinical research", inclusion (over a period arbitrarily defined from October 1, 2015 to November 1, 2015) of patients aged 75 and over with a diagnosis of fall or a related reason when they are admitted to the Emergencies Room.

During the initial consultation in the Emergency Department, documentary analysis with all the signs of seriousness of the falls stated in the report, as defined by HAS 2009:

* consequences of the fall (moderate to severe physical trauma, inability to rise from the ground and its consequences, post-fall syndrome)
* pathologies responsible for the fall
* repetitive nature of the fall (recent increase in the frequency of falls, association of more than 3 risk factors for falls, gait disorders)
* situations at risk of severe falls (proven osteoporosis, use of anticoagulant drugs, social and family isolation) Search for an anterior passage of the patient in the geriatric pathway.

Collection of the patient's care pathway following this passage to the ER:

* request for consultation or specialized geriatric care
* return home / hospitalization / Subacute care and rehabilitation

Data collected one year after the emergency department visit, based on the information available in the URQUAL and CROSSWAY databases accessible at Angers Hospital, are:

* search for passage in the geriatric pathway following the emergency consultation (external geriatric consultation, intervention of the mobile geriatric team, hospitalization in Geriatrics)
* readmission to the Emergency Department of Angers University Hospital for fall
* death Telephone call to the general practitioner one year after the initial admission, in order to search for a recurrence of fall.

This call-back makes it possible to collect data from patients readmitted for a fall in another center (clinic, hospital, etc.) or who have fallen again at home without admission to an emergency service with the aim of limiting the information and monitoring biases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Reason for emergency consultation: fall or a related cause (fracture, head trauma, etc.)

Exclusion Criteria:

* No one

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients are recruited during their passage to the Emergency Room of the University Hospital of Angers, France
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Measure of the proportion of serious fallers included in the geriatric pathway one year after passing the emergencies. | 1 year
  This outcome is assessed by the number of serious faller patients in the geriatric pathway.

SECONDARY OUTCOMES:
Measure of proportion of fallers admitted to emergencies. | baseline
  This outcome is assessed by the number of fallers admitted to emergencies.
Measure of proportion of serious fallers admitted to emergencies. | baseline
  This outcome is assessed by the number of serious fallers admitted to emergencies.
Number of severity criteria most commonly encountered in emergencies. | baseline
  This outcome is assessed by the emergencies data.
Measure of the proportion of patients who fell again within one year of admission to ER. | 1 year
  This outcome is assessed by the number of patients who fell again within one year of admission to ER.
Measure of the proportion of patients included in the geriatric pathway readmitted for fall to the ER in the following year. | 1 year
  This outcome is assessed by the number of patients included in the geriatric pathway readmitted for fall to the ER.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France